CLINICAL TRIAL: NCT03428867
Title: Phase II Studie Zur Neoadjuvanten Trimodalen Hyperthermen Radiochemotherapie Des Tief Sitzenden Rektumskarzinoms im Stadium UICC II + III
Brief Title: Register Study of the Neoadjuvanten Treatment by Patients With Rectumcarcinoma
Acronym: HT01
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Daniel Zips, Prof.Dr. med., University Hospital Tuebingen
Other Study IDs: UKT_RO_HT_01
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Feasibilitystudy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
goal of this study is to check the effecivity, feasibility and toxicity of the chemoradiotherapy and hyperthermia

DETAILED DESCRIPTION:
Radiation: 5x1,8Gy until 50,4 Gy Hyperthermia: 2x/week

Chemotherapy:

neoadjuvant= day 1-5 and day 29-33 5FU 1000mg/m2 adjuvant = 4 Cycles 5FU 500mg/m2 all 4 weeks

ELIGIBILITY:
Inclusion Criteria:

adenocarcinoma until 10 cm until ano UICC II+III 18-80 years old ECOG PS 0-2 Informed Consent

Exclusion Criteria:

cardiac insufficiency last 6 month heartattack nodal AV pressure III° hip prothesis cardiac pacemaker others contraindikations against the therapie radiation of pelvis chronic gestrointestinal desaese gestation or lactation previous radiotion pelvis previous Chemotherapie second carcinoma beside baslioma infiltation in analarea

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with rectumcarcinoma stage UICC II+III
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2012-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
remission | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Zips, Prof.Dr., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany